CLINICAL TRIAL: NCT02738892
Title: Preventing Preterm Birth in Zambia
Brief Title: Zambian Preterm Birth Prevention Study
Acronym: ZAPPS
Status: Active, not recruiting | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Global Alliance to Prevent Prematurity and Stillbirth (Unknown); Bill and Melinda Gates Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: 14-2113
Record Dates: First submitted 2016-04-06; First posted 2016-04-14 (Estimated); Last update posted 2025-06-11 (Actual); Status verified 2025-05

CONDITIONS: Pregnancy; Stillbirth; Preterm Birth
Keywords: Pregnancy; Stillbirth; Preterm birth
MeSH Terms: conditions — Stillbirth; Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, urine, vaginal, placental, and umbilical cord samples will be placed in a biorepository for later analysis to identify inflammatory markers, chemokines, cytokines, and infections contributing to parturition and preterm delivery.
Oversight: Data Monitoring Committee: No

SUMMARY:
This prospective non-intervention cohort study will enroll women in the first or early second trimester of pregnancy and follow them through delivery (or end of pregnancy) and 1 year postpartum.

Infants will also be followed until 1 year postpartum. Detailed medical and obstetrical information will be collected, as well as biological samples, in order to better elucidate the biological mechanisms leading to preterm delivery among Zambian women, in an effort to identify new strategies for prevention.

DETAILED DESCRIPTION:
After consenting to study participation, women will be asked their detailed medical and obstetrical history. Participants will be provided standard of care. Blood, urine, and vaginal specimens will also be collected for the biorepository from those who consent to participate. Participants will also be screened for depression using the Edinburgh Postnatal Depression Scale (EPDS).

Throughout the study, participants will receive education about nutrition, pregnancy health, and the signs and symptoms of complications of pregnancy, including preterm labor and preterm premature rupture of membranes. Study visits for will be scheduled at 24, 28, 32, and 36 weeks gestation, at the time of discharge from the labor and delivery ward if possible, and at 7 days, 28 days, 42 days, 6 months, and 12 months postpartum

During each study visit (i.e., at 24, 32, and 36 weeks gestation), participants will receive the routinely recommended screening and treatment. This will consist of weight, blood pressure, and symptom screening, as well as measurements of fetal growth (fundal height) and fetal well being (fetal heart rate) at each visit. Screening and treatment of common pregnancy complications will also be provided if clinically indicated. All participants will undergo maternal hemoglobin testing and urinalysis at the 24 and 32-week visits. Maternal random fasting glucose testing will be conducted at the 28-week visit to screen for gestational diabetes. Syphilis titers will be obtained at a minimum at the 36 week visit for participants seropositive at screening to monitor serologic response after treatment. HIV testing will be repeated at 28 weeks for participants uninfected at screening, and HIV Viral Load and T cell assays will be performed at the 28- and 36-week visits for any seroconverters. Participants who are HIV-infected at screening will undergo HIV Viral Load and T cell assays at 28 and 36 weeks. At 24, 28, and 36 weeks, blood, urine, oropharyngeal, and vaginal swabs will be collected. We will also collect a rectal swab at the 36-week visit. .

At the time of delivery, the study team will obtain detailed information about the clinical management of the participant's delivery, as well as the delivery outcome for both the mother and her infant(s). A urinalysis, complete blood count with differential, blood chemistry testing will be performed. We will also obtain information on interval complications and mortality. In addition, we will collect samples of the placenta, umbilical cord, and cord blood after delivery for various assessments. 4-5 drops of cord blood will be applied to designated filter paper within pre-printed circles. Newborn heel-prick samples will be collected 24-72 hours after birth or sooner if the newborn is discharged from hospital within 24 hours of delivery.

There will be four study visits during the postnatal period, at 7 days, 42 days, 6 months, and 12 months postpartum. At these visits, we will assess interval maternal or infant complications and/or mortality and measure anthropometrics. Once again, participants will receive routinely recommended screening and treatment.

Maternal hemoglobin will be measured at all post-partum visits. Urinalysis will be performed at the 42-day visit only. Maternal blood, urine, oral/pharyngeal and vaginal specimens will be collected for storage and protocol related testing at the 42-day visit. Maternal syphilis and HIV testing will be repeated at the 42-day, 6- and 12-month visits for participants who are uninfected. HIV-exposed infants will have blood collected for early infant diagnosis at the 42-day and 6- and 12-month visits; this will be done via heel prick and dried blood spot (DBS) cards requiring five drops of blood. Maternal participants will again be screened for depression using the EPDS

ELIGIBILITY:
Inclusion Criteria:

Pregnant women ≥15 years will be eligible to participate. Additionally, participants will:

1. Have a completed screening ultrasound with gestational age < 20 weeks
2. Be HIV-uninfected at enrollment (NB: prior to Protocol Version 4.0 [3 Nov 2017] enrolled both HIV-infected and uninfected women)
3. Have a singleton or twin pregnancy with fetal heart tones confirmed by ultrasound
4. Reside within Lusaka with no plans to relocate during the study follow-up period
5. Be willing to provide written, informed consent
6. Be willing to allow their infants to participate in the study

Exclusion criteria:

1. Pregnant women > 24 weeks' gestation or with screening ultrasound ≥ 16 weeks
2. Infants born to women not enrolled in the study

Ages: 15 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: The study will be conducted at Kamwala Health Centre and the University Teaching Hospital, both in Lusaka, Zambia.
Sampling Method: Non-Probability Sample
Enrollment: 9000 (Estimated)
Dates: Start 2015-08 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Preterm Birth <37 | Measured at delivery
  Proportion of deliveries occurring prior to 37 weeks gestation

SECONDARY OUTCOMES:
Preterm Birth <34 | Measured at delivery
  Proportion of deliveries occurring prior to 34 weeks gestation
Preterm Birth <28 | Measured at delivery
  Proportion of deliveries occurring prior to 28 weeks gestation
Low Birth Weight | Measured at delivery
  Proportion of newborns weighing less than 2500 grams at delivery
Very Low Birth Weight | Measured at delivery
  Proportion of newborns weighing less than 1500 grams at delivery
Preterm prelabor rupture of membranes (PPROM) | Enrollment through delivery
  Proportion of women with PPROM
Spontaneous delivery prior to 37 weeks of gestation | Enrollment through 37 weeks gestation
  Proportion of spontaneous deliveries
Spontaneous delivery prior to 34 weeks of gestation | Enrollment through 34 weeks gestation
  Proportion of spontaneous deliveries
Spontaneous delivery prior to 28 weeks of gestation | Enrollment through 28 weeks gestation
  Proportion of spontaneous deliveries
Birth weight <10th percentile for gestational age | Measured at delivery
  Proportion of newborns with birth weight < 10th percentile for gestational age
Birth weight <3rd percentile for gestational age | Measured at delivery
  Proportion of newborns with birth weight <3rd percentile for gestational age
Mother-to-child HIV transmission by 6 weeks postpartum | Delivery through 6 weeks postpartum
  Proportion of HIV positive newborns
Mother-to-child HIV transmission by 12 months postpartum | Delivery through 12 months postpartum
  Proportion of HIV positive infants
Maternal mortality | Enrollment through 12 months postpartum
  Death of a maternal participant for any reason
Fetal, neonatal, and infant mortality | Enrollment through 12 months postpartum
  Death of a fetal, neonatal, or infant participant for any reason
Infant APGAR scores | Measured at delivery
  APGAR scores at delivery

CONTACTS AND LOCATIONS:
Overall Officials: Jeff Stringer, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (2):
- Zambia (2):
  - Kamwala Health Centre, Lusaka
  - University Teaching Hospital, Lusaka

REFERENCES:
- [Background] Lawn JE, Kinney MV, Black RE, Pitt C, Cousens S, Kerber K, Corbett E, Moran AC, Morrissey CS, Oestergaard MZ. Newborn survival: a multi-country analysis of a decade of change. Health Policy Plan. 2012 Jul;27 Suppl 3:iii6-28. doi: 10.1093/heapol/czs053. PMID 22692417
- [Background] Nour NM. Premature delivery and the millennium development goal. Rev Obstet Gynecol. 2012;5(2):100-5. PMID 22866189
- [Background] Wang ML, Dorer DJ, Fleming MP, Catlin EA. Clinical outcomes of near-term infants. Pediatrics. 2004 Aug;114(2):372-6. doi: 10.1542/peds.114.2.372. PMID 15286219
- [Background] Blencowe H, Cousens S, Oestergaard MZ, Chou D, Moller AB, Narwal R, Adler A, Vera Garcia C, Rohde S, Say L, Lawn JE. National, regional, and worldwide estimates of preterm birth rates in the year 2010 with time trends since 1990 for selected countries: a systematic analysis and implications. Lancet. 2012 Jun 9;379(9832):2162-72. doi: 10.1016/S0140-6736(12)60820-4. PMID 22682464
- [Background] March of Dimes P, Save the Children, WHO. Born Too Soon: The Global Action Report on Preterm Birth. In. Edited by Eds CP Howson MK, JE Lawn. Geneva: World Health Organization; 2012.
- [Background] Goldenberg RL, Culhane JF, Iams JD, Romero R. Epidemiology and causes of preterm birth. Lancet. 2008 Jan 5;371(9606):75-84. doi: 10.1016/S0140-6736(08)60074-4. PMID 18177778
- [Background] Oliver RS, Lamont RF. Infection and antibiotics in the aetiology, prediction and prevention of preterm birth. J Obstet Gynaecol. 2013 Nov;33(8):768-75. doi: 10.3109/01443615.2013.842963. PMID 24219711
- [Background] Gotsch F, Gotsch F, Romero R, Erez O, Vaisbuch E, Kusanovic JP, Mazaki-Tovi S, Kim SK, Hassan S, Yeo L. The preterm parturition syndrome and its implications for understanding the biology, risk assessment, diagnosis, treatment and prevention of preterm birth. J Matern Fetal Neonatal Med. 2009;22 Suppl 2:5-23. doi: 10.1080/14767050902860690. No abstract available. PMID 19951079
- [Background] Lawn JE, Cousens S, Zupan J; Lancet Neonatal Survival Steering Team. 4 million neonatal deaths: when? Where? Why? Lancet. 2005 Mar 5-11;365(9462):891-900. doi: 10.1016/S0140-6736(05)71048-5. PMID 15752534
- [Background] Iams JD. Clinical practice. Prevention of preterm parturition. N Engl J Med. 2014 Jan 16;370(3):254-61. doi: 10.1056/NEJMcp1103640. No abstract available. PMID 24428470
- [Background] Muglia LJ, Katz M. The enigma of spontaneous preterm birth. N Engl J Med. 2010 Feb 11;362(6):529-35. doi: 10.1056/NEJMra0904308. No abstract available. PMID 20147718
- [Background] Kim CJ, Romero R, Kusanovic JP, Yoo W, Dong Z, Topping V, Gotsch F, Yoon BH, Chi JG, Kim JS. The frequency, clinical significance, and pathological features of chronic chorioamnionitis: a lesion associated with spontaneous preterm birth. Mod Pathol. 2010 Jul;23(7):1000-11. doi: 10.1038/modpathol.2010.73. Epub 2010 Mar 26. PMID 20348884
- [Background] Myatt L, Eschenbach DA, Lye SJ, Mesiano S, Murtha AP, Williams SM, Pennell CE; International Preterm Birth Collaborative Pathways and Systems Biology Working Groups. A standardized template for clinical studies in preterm birth. Reprod Sci. 2012 May;19(5):474-82. doi: 10.1177/1933719111426602. Epub 2012 Feb 16. PMID 22344727
- [Background] Romero R, Espinoza J, Kusanovic JP, Gotsch F, Hassan S, Erez O, Chaiworapongsa T, Mazor M. The preterm parturition syndrome. BJOG. 2006 Dec;113 Suppl 3(Suppl 3):17-42. doi: 10.1111/j.1471-0528.2006.01120.x. PMID 17206962
- [Background] Romero R, Espinoza J, Gotsch F, Kusanovic JP, Friel LA, Erez O, Mazaki-Tovi S, Than NG, Hassan S, Tromp G. The use of high-dimensional biology (genomics, transcriptomics, proteomics, and metabolomics) to understand the preterm parturition syndrome. BJOG. 2006 Dec;113 Suppl 3(Suppl 3):118-35. doi: 10.1111/j.1471-0528.2006.01150.x. PMID 17206980
- [Background] Liong S, Di Quinzio MK, Fleming G, Permezel M, Rice GE, Georgiou HM. Prediction of spontaneous preterm labour in at-risk pregnant women. Reproduction. 2013 Aug 21;146(4):335-45. doi: 10.1530/REP-13-0175. Print 2013 Oct. PMID 23858477
- [Background] Cox JL, Holden JM, Sagovsky R. Detection of postnatal depression. Development of the 10-item Edinburgh Postnatal Depression Scale. Br J Psychiatry. 1987 Jun;150:782-6. doi: 10.1192/bjp.150.6.782. PMID 3651732
- [Background] Wisner KL, Parry BL, Piontek CM. Clinical practice. Postpartum depression. N Engl J Med. 2002 Jul 18;347(3):194-9. doi: 10.1056/NEJMcp011542. No abstract available. PMID 12124409
- [Background] Aleman A, Cafferata ML, Gibbons L, Althabe F, Ortiz J, Sandoval X, Padilla-Raygoza N, Belizan JM. Use of antenatal corticosteroids for preterm birth in Latin America: providers knowledge, attitudes and practices. Reprod Health. 2013 Jan 29;10:4. doi: 10.1186/1742-4755-10-4. PMID 23360713
- [Background] Crowley P. Prophylactic corticosteroids for preterm birth. Cochrane Database Syst Rev. 2000;(2):CD000065. doi: 10.1002/14651858.CD000065. PMID 10796110
- [Derived] Appiagyei A, Vwalika B, Spelke MB, Conner MG, Mabula-Bwalya CM, Kasaro MP, Honart AW, Kumwenda A, Stringer EM, Stringer JSA, Price JT. Maternal mid-upper arm circumference to predict small for gestational age: Findings in a Zambian cohort. Int J Gynaecol Obstet. 2023 May;161(2):462-469. doi: 10.1002/ijgo.14517. Epub 2022 Oct 31. PMID 36263879
- [Derived] Price JT, Vwalika B, Edwards JK, Cole SR, Kasaro MP, Rittenhouse KJ, Kumwenda A, Lubeya MK, Stringer JSA. Maternal HIV Infection and Spontaneous Versus Provider-Initiated Preterm Birth in an Urban Zambian Cohort. J Acquir Immune Defic Syndr. 2021 Jun 1;87(2):860-868. doi: 10.1097/QAI.0000000000002654. PMID 33587508
- [Derived] Rittenhouse KJ, Mwape H, Nelson JAE, Mwale J, Chipili G, Price JT, Hudgens M, Stringer EM, De Paris K, Vwalika B, Stringer JSA. Maternal HIV, antiretroviral timing, and spontaneous preterm birth in an urban Zambian cohort: the role of local and systemic inflammation. AIDS. 2021 Mar 15;35(4):555-565. doi: 10.1097/QAD.0000000000002808. PMID 33394679
- [Derived] Rittenhouse KJ, Vwalika B, Keil A, Winston J, Stoner M, Price JT, Kapasa M, Mubambe M, Banda V, Muunga W, Stringer JSA. Improving preterm newborn identification in low-resource settings with machine learning. PLoS One. 2019 Feb 27;14(2):e0198919. doi: 10.1371/journal.pone.0198919. eCollection 2019. PMID 30811399
- See also: University of North Carolina website — http://www.unc.edu